CLINICAL TRIAL: NCT00879268
Title: Phase 1 Study of Liver Machine Preservation With Vasosol Solution
Brief Title: Vasosol Organ Perfusion Solution and Medtronic Portable Bypass System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polyak, Maximilian (Individual)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Dr. James V. Guarrera, Columbia University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G030132
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Liver Transplantation; Organ Preservation
Keywords: Liver Transplantation; Organ Preservation; Liver Preservation; Machine Perfusion; Vasosol; Machine Preservation

INTERVENTIONS:
Device: Vasosol Organ Perfusion Solution and Medtronic Portable Bypass System — Utilization of Vasosol with Medtronic System for Machine Preservation of the Liver for Liver Transplantation
  Other Names: Vasosol Solution; Medtronic Portable Bypass System

SUMMARY:
This is a pilot trial of centrifugal machine preservation of donor livers for transplantation using a novel preservation solution.

ELIGIBILITY:
Inclusion Criteria:

* Primary/ Solitary Liver Transplant
* Lab MELD<35
* Donor age <65

Exclusion Criteria:

* Donor Liver > 30% Macrosteatosis
* DCD donor liver
* Multi-organ Recipient
* Recipient in ICU
* Retransplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V. Guarrera, M.D., Principal Investigator — Columbia University